CLINICAL TRIAL: NCT03940846
Title: CT-based Radiomic Signature Can Identify Adenocarcinoma Lung Tumor Histology
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Maastricht University (Other)
Collaborators: University of California, San Francisco (Other); Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: LHist
Record Dates: First submitted 2019-05-06; First posted 2019-05-07 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2019-04

CONDITIONS: Nonsmall Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Maastro (Lung1): Open source dataset available at TCIA.org. The cohort includes CT scans of 422 patients diagnosed with NSCLC.
  Interventions: Diagnostic Test: Virtual biopsy
- UCSF: A cohort of patients diagnosed with NSCLC at UCSF medical center. It includes CT scans of 165 patients.
  Interventions: Diagnostic Test: Virtual biopsy
- Radboud: A cohort of patients diagnosed with NSCLC at Radboud medical center. It includes CT scans of 255 patients.
  Interventions: Diagnostic Test: Virtual biopsy
- Stanford: Open source dataset available at TCIA.org. The cohort includes CT scans of 211 patients diagnosed with NSCLC.
  Interventions: Diagnostic Test: Virtual biopsy

INTERVENTIONS:
Diagnostic Test: Virtual biopsy — Radiomics -the high throughput extraction of quantitative features from medical imaging- extract features that might potentially decode biologic tumor information, which might ultimately reduce the need to use invasive procedure, such as tissue biopsy.
  Other Names: Radiomics-based histology prediction

SUMMARY:
Lung cancer remains the leading cause of cancer related mortality worldwide, with more than 1.5 million related deaths annually. Lung cancer is divided into two main groups: Small Cell Lung Carcinoma (SCLC) and Non-Small Cell Lung Carcinoma (NSCLC), with prevalence of ~20% and 80% respectively. NSCLC is further subdivided into adenocarcinoma (the most common), squamous cell carcinoma (SCC), and large cell carcinoma. Furthermore, each subtype is likely to have specific mutations, which could be targeted for treatment.

Medical imaging and radiomics feature extraction represent a candidate alternative to conventional tissue biopsy, a theory that is investigated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Availability of diagnostic non-contrast enhanced CT scan.
* Availability of histologic tumor analysis results

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with NSCLC, who further underwent tissue biopsy to determine tumor histology.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Lung histology | December 2019
  Is the tumor under investigation an adenocarcinoma of the lung?

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided